CLINICAL TRIAL: NCT06330805
Title: A Comparison of Orgovyx (Relugolix) vs Eligard (Leuprolide) on Cardiovascular Function and Biomarkers During Standard of Care Combined ADT (Androgen Deprivation Therapy)-Radiation for Prostate Cancer
Brief Title: Effects of Relugolix vs Leuprolide on Cardiac Function in Patients With Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry); Myovant Sciences GmbH (Industry); Sumitomo Pharmaceuticals America (Industry)
Responsible Party: Principal Investigator, Shang-Jui Wang, MD, PhD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-23069; NCI-2024-00705 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-03-02; First posted 2024-03-26 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Prostate Adenocarcinoma; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Contrast Media; Leuprolide; Magnetic Resonance Spectroscopy; Exercise Test; relugolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (leuprolide) (Experimental): Patients receive definitive therapy for prostate cancer with ADT (leuprolide via injection once every 3 months, for a total of 6 months) in the absence of disease progression or unacceptable toxicity and definitive radiotherapy within 90 days of starting ADT. Patients receive gadolinium-based contrast intravenously (IV) and undergo exercise-stress cardiac MRI perfusion and comprehensive exercise physiology testing before starting ADT and at 6 months after starting ADT. Patients also undergo blood and urine sample collection throughout the study, as well as completion of quality-of-life questionnaires.
  Interventions: Procedure: Biospecimen Collection; Other: Contrast Agent; Drug: Leuprolide; Procedure: Magnetic Resonance Imaging; Other: Physical Performance Testing
- Arm 2 (relugolix) (Experimental): Patients receive definitive therapy for prostate cancer with ADT (relugolix orally once daily for a total of 6 months) in the absence of disease progression or unacceptable toxicity and definitive radiotherapy within 90 days of starting ADT. Patients receive gadolinium-based contrast intravenously (IV) and undergo exercise-stress cardiac MRI perfusion and comprehensive exercise physiology testing before starting ADT and at 6 months after starting ADT. Patients also undergo blood and urine sample collection throughout the study, as well as completion of quality-of-life questionnaires.
  Interventions: Procedure: Biospecimen Collection; Other: Contrast Agent; Procedure: Magnetic Resonance Imaging; Other: Physical Performance Testing; Drug: Relugolix

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Contrast Agent — Given IV
  Other Names: Contrast; Contrast Drugs; contrast material; Contrast Medium
Drug: Leuprolide — Given injection
  Other Names: Leuprorelin
  Arms: Arm 1 (leuprolide)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Physical Performance Testing — Undergo functional fitness tests
  Other Names: Physical Fitness Testing; Physical Function Testing
Drug: Relugolix — Given PO
  Other Names: N-(4-(1-((2,6-Difluorophenyl)methyl)-5-((dimethylamino)methyl)-1,2,3,4-tetrahydro-3-(6-methoxy-3-pyridazinyl)-2,4-dioxothieno(2,3-d)pyrimidin-6-yl)phenyl)-N'-methoxyurea; Orgovyx; Relumina; TAK 385; TAK-385
  Arms: Arm 2 (relugolix)

SUMMARY:
This phase II trial compares the effect of relugolix to leuprolide on cardiac function and performance in patients with prostate cancer. Androgen deprivation therapy (ADT) has been a key component for the treatment of advanced prostate cancer for decades. The term androgen deprivation therapy means lowering a man's testosterone. Long-term studies show that ADT may contribute to a detriment to cardiac health and predisposes men to developing cardiac diseases. Recent studies suggest that men taking relugolix for treatment of prostate cancer may have a lower risk of developing cardiovascular problems, but more studies are needed to understand this observation, and there are currently no studies reporting the direct impact of ADT (relugolix, versus the more-commonly used leuprolide) on cardiac function and outcomes.

Participants will receive definitive radiotherapy for unfavorable intermediate risk prostate cancer and 6-month ADT (either relugolix or leuprolide). In addition, participants will undergo the following:

1. Comprehensive cardiac and exercise testing before and after starting ADT
2. Completion of quality-of-life questionnaires at specific intervals during the study period
3. Provide blood samples at specific intervals during the study period to test for changes in steroid levels and certain biomarkers

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To quantify the physiologic alterations in cardiopulmonary function in men receiving 6-month relugolix verse (vs.) 6-month leuprolide with definitive radiation therapy (RT) for unfavorable intermediate risk (UIR) clinically localized prostate cancer (PCa).

II. Cardiopulmonary and cardiac measures obtained from: 1) exercise stress cardiac magnetic resonance imaging (MRI) perfusion, and 2) maximal rate of oxygen consumption (VO2), include myocardial perfusion reserve index (MPRI), contractile reserve, myocardial longitudinal relaxation time (T1) signal, longitudinal strain, circumferential strain, VO2 maximum (max), and metabolic equivalents of exercise capacity (METs).

SECONDARY OBJECTIVES:

I. To quantify the impact of 6-month relugolix vs. leuprolide with definitive RT for UIR PCa on quality of life (QoL) using Expanded Cancer Index Composite (EPIC)-26, European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30), European (Euro) Qol-5-Dimension 5-level (EQ-5D-5L), and Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue (Short Form 8a) patient-reported outcome surveys, or similar tests.

II. To quantify the impact of 6-month relugolix vs. leuprolide on composite functional tests of strength and balance using three tests: 1) Timed Up-and-Go, 2) 10-meter walk time, and 3) grip strength.

III. To analyze body composition changes in response to 6-month relugolix vs. leuprolide by using abdominal computed tomography (CT) or magnetic resonance imaging (MRI) to quantitate abdominal/visceral fat and lean muscle mass with utilization of SliceOmatic software.

EXPLORATORY OBJECTIVES:

I. To compare changes in serum steroid profiles (panel of 17 steroid hormone metabolites, Ohio State University Comprehensive Cancer Center [OSUCCC Pharmacoanalytic Shared Resource [PhASR]) before, during and after 6-month relugolix vs. 6-month leuprolide with definitive RT for UIR PCa.

II. To compare changes in cardiometabolic biomarkers in the following three categories: 1) glycemic control parameters (fasting glucose, fasting insulin, and connecting [C]-peptide), 2) lipid profiles (total cholesterol, triglyceride, low-density lipoprotein [LDL], high-density lipoprotein [HDL], and leptin/adiponectin ratio), 3) markers of the obesity-associated low-grade chronic inflammatory state (CRP, TGF-beta, and IL-6, and novel related immunoregulators), and targeted or non- targeted metabolomics or proteomics (by OSUCCC NPASR and PSR) depending on procurement of additional funds.

III. To compare the time course of recovery for hormonal and cardiometabolic markers after completion of 6-month relugolix vs. 6-month leuprolide with definitive RT for UIR PCa.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive definitive therapy for prostate cancer with ADT (leuprolide via injection once every 3 months, for a total of 6 months) in the absence of disease progression or unacceptable toxicity and definitive radiotherapy within 90 days of starting ADT. Patients receive gadolinium-based contrast intravenously (IV) and undergo exercise-stress cardiac MRI perfusion and comprehensive exercise physiology testing before starting ADT and at 6 months after starting ADT. Patients also undergo blood and urine sample collection throughout the study, as well as completion of quality-of-life questionnaires.

ARM 2: Patients receive definitive therapy for prostate cancer with ADT (relugolix orally once daily for a total of 6 months) in the absence of disease progression or unacceptable toxicity and definitive radiotherapy within 90 days of starting ADT. Patients receive gadolinium-based contrast intravenously (IV) and undergo exercise-stress cardiac MRI perfusion and comprehensive exercise physiology testing before starting ADT and at 6 months after starting ADT. Patients also undergo blood and urine sample collection throughout the study, as well as completion of quality-of-life questionnaires.

After completion of study treatment, patients are followed up at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of adenocarcinoma of the prostate within 270 days prior to registration.
* Unfavorable intermediate risk prostate cancer, defined as having ALL the following bulleted criteria:

  * Has at least one intermediate risk factor (IRF):

    * Prostate-specific antigen (PSA) 10-20 ng/mL
    * Clinical stage tumor (T)2b-c (digital rectal exam [DRE] and/or imaging) by American Joint Committee on Cancer (AJCC) 8th edition
    * Gleason Score 7 (Gleason 3+4 or 4+3 [International Society of Urological Pathology [ISUP] grade group 2-3])
  * Has one or more of the following "unfavorable" intermediate-risk designators:

    * > 1 IRF
    * Gleason 4+3=7 (ISUP grade group 3)
    * ≥ 50% of biopsy cores positive

      * Biopsies may include "sextant" sampling of right/left regions of the prostate, often labeled base, mid-gland and apex. All such "sextant" biopsy cores should be counted. Men may also undergo "targeted" sampling of prostate lesions (guided by MRI, ultrasound or other approaches). A targeted lesion that is biopsied more than once and demonstrates cancer (regardless of number of targeted cores involved) should count as a single additional positive core sampled and positive. In cases of uncertainty, count the biopsy sampling as sextant core(s).
    * Absence of high-risk features
* Appropriate stage based on the following diagnostic workup:

  * History/physical examination within 120 days prior to registration
  * Negative bone imaging (M0) with Tc-99m bone scan or fluciclovine (18F) sodium fluoride (NaF) positron emission tomography (PET) within 120 days prior to registration
  * Clinically negative lymph nodes (N0) as established by conventional imaging (pelvic +/- abdominal CT or MRI), within 120 days prior to registration (lymph nodes equivocal or questionable by imaging are eligible if the nodes are ≤ 1.0 cm in short axis and/or if biopsy is negative)
  * Prostate specific membrane antigen (PSMA) or fluciclovine PET negative for nodal or distant metastatic disease is an acceptable substitute for the above bone and pelvic imaging
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1 within 120 days prior to registration.
* Non-castrate testosterone level (> 50 ng/dL) within 120 days prior to registration.
* Absolute neutrophil ≥ 1,000 cells/mm^3 (within 120 days prior to registration)
* Hemoglobin ≥ 10 g/dL (within 120 days prior to registration)
* Platelet count ≥ 100,000 cells/mm^3 (within 120 days prior to registration)
* Creatinine clearance (CrCl) ≥ 30 mL/min estimated by Cockcroft-Gault Equation (within 120 days prior to registration)

  * For African American patients, CrCl ≥ 30 mL/min is estimated by the alternative formula that takes race into account
* Total bilirubin: 1.5 ≤ institutional upper limit of normal (ULN) (within 120 days prior to registration)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT)(serum glutamic-pyruvic transaminase [SGPT]) ≤ 2.5 × institutional ULN (within 120 days prior to registration)
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. Note: HIV testing is not required for eligibility for this protocol.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.

Note: Known positive test for hepatitis B virus surface antigen (HBV sAg) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy. Patients who are immune to hepatitis B (anti-Hepatitis B surface antibody positive) are eligible (e.g. patients immunized against hepatitis B).

* For patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.

  * Note: Known positive test for hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy.
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information.

Exclusion Criteria:

* Previous radical surgery (prostatectomy) or any form of curative-intent ablation whether focal or whole-gland (e.g., cryosurgery, High-intensity focused ultrasound (HIFU), laser thermal ablation, etc.) for prostate cancer.
* Definitive clinical or radiologic evidence of metastatic disease (M1).
* Prior invasive malignancy (except non-melanomatous skin cancer) or hematologic malignancy unless disease free for a minimum of 3 years.
* Prior radiotherapy to the prostate/pelvis region that would result in overlap of radiation therapy fields.
* Previous bilateral orchiectomy.
* Previous hormonal therapy, such as luteinizing hormone-releasing hormone (LHRH) agonists (e.g., leuprolide, goserelin, buserelin, triptorelin) or LHRH antagonist (e.g. degarelix), anti-androgens (e.g., flutamide, bicalutamide, cyproterone acetate). ADT started prior to study registration is not allowed.
* Prior use of 5-alpha-reductase inhibitors is allowed; however, it must be stopped ≥ 30 days prior to the pre-registration PSA measure for determining enrollment eligibility.
* Prior testosterone replacement therapy is allowed; however, any replacement therapy must be stopped for at least 1 year prior to registration.
* Severe, active co-morbidity defined as follows:

  * Current/uncontrolled angina or arrhythmias
  * New York Heart Association Functional Classification II-IV (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification.)
  * History of any condition that in the opinion of the investigator, would preclude participation in this study
* Patients with significant obstructive urinary symptoms that are suspected to be secondary to prostate cancer and/or benign prostatic hypertrophy.
* Disabilities that prevent performing moderate intensity exercise test with exercise (treadmill) stress test and muscle function tests (walking/gait assessments and grip strength).
* Patients unable to tolerate MRI (e.g. claustrophobia), has contraindications to MRI (e.g. metals and implants incompatible with MRI), body habitus preventing MRI scanning, or allergy to gadolinium-based contrast.
* Significant uncontrolled gastrointestinal (e.g. Crohn's disease, ulcerative colitis) or metabolic disease (e.g. diabetes, hyperlipidemia).
* Active inflammatory or immune-related disease treated with steroids or immunosuppressive agents.
* Inability to swallow oral pills.
* High risk features, which includes any of the following:

  * Gleason 8-10 [ISUP grade group 4-5]
  * PSA>20
  * cT3-4 by digital exam OR gross extra-prostatic extension on imaging [indeterminate MRI evidence will not count and the patient will be eligible]

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Physiologic alterations in cardiopulmonary function - Myocardial perfusion | Up to 6 months
  We will measure the difference in myocardial perfusion with exercise stress-rest cardiac MRI before and after ADT (leuprolide vs. relugolix).
Physiologic alterations in cardiopulmonary function - Maximal rate of oxygen consumption | Up to 6 months
  We will measure the difference in VO2 Max before and after ADT (leuprolide vs. relugolix).

SECONDARY OUTCOMES:
Quality of life using EPIC-26 | Up to 6 months
  Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale. Overall, higher scores across the EPIC domains represent better QoL.
Quality of life using EORTC QLQ-C30 | Up to 6 months
  All of the scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning.
Quality of life using European (Euro) Qol-5-Dimension 5-level (EQ-5D-5L) | Up to 6 months
  This validated utility assessment instrument evaluates 5-dimensions (5D) of function, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each graded on 5 levels (ranging from 1 [no problem] to 5 [extreme problems]). The 5D index score is transformed into a utility score between 0 and 1. The sixth item is a visual analogue scale for overall health perceived by the patient. A lower score represents better health.
Quality of life using PROMIS | Up to 6 months
  A 5-point Likert scale from 1 (never/not at all) to 5 (almost always/very much) with a recall period of last 7 days. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean.
Functional tests of strength and balance using Timed Up-and-Go | Up to 6 months
  Participants will be instructed to stand up from an armchair (seat height of 45 cm), walk at a comfortable pace to a line on the floor 3 meters away, turn, return to the chair and sit down again. A stopwatch is used to time the performance (in seconds).
Functional tests of strength and balance using 10-meter walk time | Up to 6 months
  Gait speed will be measured using a standardized 10-m course.
Functional tests of strength and balance using Grip strength | Up to 6 months
  A validated biomarker of overall strength and muscle mass. Patients will perform 3 trials with each hand, alternating hands between trials, with the maximum score for each hand being recorded.
Changes in body composition | Up to 6 months
  Abdominal CT/MRI to quantitate abdominal/visceral fat and lean muscle mass with utilization of image analysis software.

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Jui Wang, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu